CLINICAL TRIAL: NCT06928584
Title: Multicenter, Randomized, Phase II Trial of Neoadjuvant Hypofractionated Radiotherapy Plus Immunotherapy and First-line Therapy Versus Conventional Radiotherapy Plus First-line Therapy in pMMR Locally Recurrent Rectal Cancer (TORCH-R2)
Brief Title: Hypofractionated Radiotherapy Plus Immunotherapy Versus Conventional Radiotherapy in Locally Recurrent Rectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhen Zhang, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDRT-2024-416-3970
Record Dates: First submitted 2025-04-08; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Locally Recurrent Rectal Cancer
MeSH Terms: interventions — Capecitabine; Fluorouracil; Leucovorin; Oxaliplatin; Irinotecan; Cetuximab; Bevacizumab; Radiation Dose Hypofractionation; spartalizumab; sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional radiotherapy arm (Active Comparator): Conventional radiotherapy (50Gy/25Fx irradiation or 39Gy/30Fx bid reirradiation) and investigator's choice of first-line chemotherapy +/- target therapy.
  Interventions: Radiation: Conventional Radiotherapy; Drug: Capecitabine; Drug: 5-fluorouracil; Drug: folinic acid; Drug: Oxaliplatin; Drug: Irinotecan; Drug: Cetuximab; Drug: Bevacizumab
- Hypofractionated radiotherapy plus Immunotherapy arm (Experimental): Hypofractionated radiotherapy (25-40Gy/5Fx irradiation or 15-30Gy/5Fx reirradiation), 18 weeks sintilimab and investigator's choice of first-line chemotherapy +/- target therapy.
  Interventions: Drug: Capecitabine; Drug: 5-fluorouracil; Drug: folinic acid; Drug: Oxaliplatin; Drug: Irinotecan; Drug: Cetuximab; Drug: Bevacizumab; Radiation: Hypofractionated radiotherapy; Drug: PD-1 antibody

INTERVENTIONS:
Radiation: Conventional Radiotherapy — 50Gy/25Fx irradiation or 39Gy/30Fx bid reirradiation (previous pelvic radiation)
  Arms: Conventional radiotherapy arm
Drug: Capecitabine — 1000mg/m2 d1-14 q3w
Drug: 5-fluorouracil — 400 mg/m2 (bolus) and 2400 mg/m2 (continuous infusion for 48hr)
Drug: folinic acid — 400 mg/m2 q2w
Drug: Oxaliplatin — 130 mg/m² q3w or 85 mg/m² q2w
Drug: Irinotecan — 180 mg/m² q2w and 200 mg/m² q3w
Drug: Cetuximab — 500 mg/m² q2w
Drug: Bevacizumab — 5 mg/kg q2w or 7.5mg/kg q3w
Radiation: Hypofractionated radiotherapy — 25-40Gy/5Fx irradiation or 15-30Gy/5Fx reirradiation (previous pelvic radiation)
  Arms: Hypofractionated radiotherapy plus Immunotherapy arm
Drug: PD-1 antibody — 200mg IV q3w
  Other Names: Sintilimab
  Arms: Hypofractionated radiotherapy plus Immunotherapy arm

SUMMARY:
TORCH-R2 is a prospective, multicenter, randomized, phase II clinical trial. Patients aged 18 years or older with pelvic recurrence rectal cancer without synchronous distant metastases or recent chemo- and/or radiotherapy treatment, Eastern Cooperative Oncology Group performance status of 0-1will be enrolled . Patients will be randomized to receive either hypofractionated radiotherapy (25-40Gy/5Fx irradiation or 15-30Gy/5Fx reirradiation), 18 weeks sintilimab and investigator's choice of first-line chemotherapy +/- target therapy (experimental arm), or conventional radiotherapy (50Gy/25Fx irradiation or 39Gy/30Fx bid reirradiation) and chemotherapy +/- target therapy (control arm). Patiens will be restaged and followed by multidisciplinary team (MDT) for decision: radical surgery, sustained systerm+/- local treatment of non resection.

The primary endpoint was progression-free survival. Secondary endpoints were objective response rate (ORR), complete response rate, R0 resection rate, duration of response (DOR), overall survival (OS), and safety and tolerability of the treatment.

ELIGIBILITY:
Inclusion Criteria:

Patient is 18-75 years. ECOG performance status 0-1. MRI/enhanced CT confirmed pelvic recurrence. Without synchronous distant metastases. No prior radiotherapy within 6 month. No prior first-line chemotherapy. Has an investigator determined life expectancy of at least 24 weeks. Demonstrate adequate organ function. Non pregnant or lactating patients. Fully informed and willing to provide written informed consent for the trial.

Exclusion Criteria:

Neutrophil< 1.5×109/L, PLT< 100×109/L (PLT< 80×109/L in patients with livermetastasis), or Hb< 90 g/L.

TBIL > 1.5 ULN, or TBIL > 2.5 ULN in patients with liver metastasis. AST or ALT > 2.5 ULN, or ALT and/or AST > 5 ULN in patients with liver metastasis.

Cr > 1.5 ULN, or creatinine clearance< 50 mL/min (calculated according to Cockcroft Gault formula).

APTT > 1.5 ULN, PT > 1.5 ULN (subject to the normal value of the clinical trial research center).

Serious electrolyte abnormalities. Urinary protein ≥ 2+, or 24-h urine protein ≥1.0 g/24 h. Uncontrolled hypertension: SBP >140 mmHg or DBP > 90 mmHg. A history of arterial thrombosis or deep vein thrombosis within 6 months; a history of bleeding or evidence of bleeding tendency within 2 months.

A history of heart disease within 6 months. Uncontrolled malignant pleural effusion, ascites, or pericardial effusion. History of checkpoint inhibitor therapy. The presence of a clinically detectable second primary malignancy, or history of other malignancies within 5 years.

A history of liver disease including, but not limited to, HBV infection or HBV DNA positive (≥1×104/mL), HCV infection or HCV DNA positive (≥1×103/mL), and liver cirrhosis.

Pregnant or lactating women or women who may be pregnant have a positive pregnancy test before the first medication, or the female participants themselves and their partners who were unwilling to implement strict contraception during the study period.

The investigator considers that the subject is not suitable to participate in this clinical study due to any clinical or laboratory abnormalities or compliance problems.

Serious mental abnormalities. The diameter of brain metastasis is greater than 3 cm or the total volume is greater than 30 cc. Clinical or radiological evidence of spinal cord compression, or tumors within 3 mm of the spinal cord on MRI.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2030-03-10 (Estimated); Study Completion 2030-03-10 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | up to 3 years
  time from the date of start treatment until disease progression or censored at last follow-up or death.

SECONDARY OUTCOMES:
Objective response rate (ORR) | up to 1 year
  the proportion of patients with the best response of confirmed complete or partial response according to RECIST 1.1, as assessed by the investigator.
Complete response rate | up to 1 year
  the proportion of patients with the best response of confirmed complete response according to RECIST 1.1, as assessed by the investigator.
R0 resection rate | up to 1 year
  the proportion of patients who achieve R0 resection of pelvic recurrent tumour after therapy.
Duration of response (DOR) | up to 3 years
  time from the first documented pelvic objective response to pelvic or extrapelvic disease progression in patients with confirmed response.
Overall Survival | up to 3 years
  from the date of start treatment until the date of death from any cause or censored at last follow-up.
Safety and tolerability | up to 1 year
  proportion of patients with treatment-related acute toxicities as assessed by NCI CTCAE v5.0, from treatment initiation until 90 days upon completion of immunotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Zhang, MD PhD, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China